CLINICAL TRIAL: NCT05960071
Title: Effects of Alveolar Recruitment Strategies on Arterial Oxygenation and Postoperative Inflammatory Response During Laparoscopic Bariatric Surgery: A Randomised Control Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0305904
Record Dates: First submitted 2023-07-18; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-06

CONDITIONS: Bariatric Surgery Candidate
Keywords: bariatric; atelectasis; alveolar recruitment
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: 60 adult obese patients (18-65 years), with American Society of Anaesthesiologists physical Status classification 1-2, enrolled in 2 groups; Group S: received protective lung strategy with recruitment manoeuvre (RM) every 30 minutes and steady PEEP (10) cm H2o in between RM till end of surgery. Group D: received protective lung strategy with recruitment manoeuvre (RM) every 30 minutes and decreasing PEEP (15, 10, and 5) cm H20 (10 minutes for each level) in between RM till end of surgery.
Who Masked: Participant
Masking Description: single blinded study where participants were not aware to the study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Active Comparator): patients received protective lung strategy with recruitment manoeuvre (RM) every 30 minutes and steady PEEP (10) cm H2O in between RM till end of surgery.
  Interventions: Procedure: protective lung strategy with recruitment manoeuvre (RM) - steady PEEP
- Group D (Active Comparator): patients received protective lung strategy with recruitment manoeuvre (RM) every 30 minutes and decreasing PEEP (15, 10, and 5) cm H20 (10 minutes for each level) in between RM till end of surgery.
  Interventions: Procedure: protective lung strategy with recruitment manoeuvre (RM) - decreasing PEEP

INTERVENTIONS:
Procedure: protective lung strategy with recruitment manoeuvre (RM) - steady PEEP — protective lung strategy with recruitment manoeuvre (RM) every 30 minutes and steady PEEP (10) cm H2o in between RM till end of surgery.
  Arms: Group S
Procedure: protective lung strategy with recruitment manoeuvre (RM) - decreasing PEEP — protective lung strategy with recruitment manoeuvre (RM) every 30 minutes and decreasing PEEP (15, 10, and 5) cm H20 (10 minutes for each level) in between RM till end of surgery.
  Arms: Group D

SUMMARY:
even though the advancement of ambulatory bariatric surgeries, yet the precise spot of recruitment manoeuvres as a secure and efficient approach to enhance the respiratory efficacy of obese patients is still obscured. Previous research have extensively focused their attention towards alveolar recruitment with various positive end-expiratory pressure (PEEP) levels to alleviate anaesthesia induced pulmonary collapse and enhance arterial oxygenation.

Patients and methods: a prospective randomized study involved 60 adult obese patients (18-65 years), with American Society of Anaesthesiologists physical Status classification 1-2, enrolled in 2 groups; Group S: received protective lung strategy with recruitment manoeuvre (RM) every 30 minutes and steady PEEP (10) cm H2o in between RM till end of surgery. Group D: received protective lung strategy with recruitment manoeuvre (RM) every 30 minutes and decreasing PEEP (15, 10, and 5) cm H20 (10 minutes for each level) in between RM till end of surgery.

DETAILED DESCRIPTION:
* Atelectasis arises shortly following onset of anaesthesia even among a healthy volunteer, and is closely correlated to escalation of intrapulmonary hypoxemia and inevitable gas exchange derangement .
* sixty adult obese patients (body mass index more than 35 kg/m2), of both sexes, aged from 18-65 years old, with American Society of Anaesthesiologists physical Status classification scores of 1-2, scheduled for laparoscopic bariatric procedures. Exclusion criteria were patients refusal, history of significant pulmonary disease (obstructive or restrictive), previous pneumothorax, significant cardiac dysfunction (arrhythmias ± unstable haemodynamics, left ventricular ejection fraction < 40%), difficult intubation as well as those suffering from significant hepatic or renal impairment. Furthermore, patients developed episodes of hemodynamic instability (like desaturation (Sp02< 90 %) or mean blood pressure (MAP) < 60 mmHg) during recruitment manoeuvre were omitted from the study.
* Subjects were randomly assigned -via closed envelopes technique opened immediately before induction- into 2 equal groups (n=30 each) to receive 1 of the following ventilatory regimens:

  * Group S: patients received protective lung strategy with recruitment manoeuvre (RM) every 30 minutes and steady PEEP (10) cm H2o in between RM till end of surgery.
  * Group D: patients received protective lung strategy with recruitment manoeuvre (RM) every 30 minutes and decreasing PEEP (15, 10, and 5) cm H20 (10 minutes for each level) in between RM till end of surgery.
* Anaesthesia was induced with lidocaine (1mg/kg) followed by (1.5 - 2 mg/kg) propofol (ideal body weight) and (1-1.5 μg/kg) fentanyl. Endotracheal intubation was accomplished with rocuronium (1mg/kg) and a suitable sized tube (8.0 ID). Anaesthesia was maintained with sevoflurane (1-2 %) with (50 %) oxygen in air. Neuromuscular block was continued with rocuronium boluses monitored by train-of four along with additional doses of opioids given as required to achieve a suitable clinical depth of anaesthesia. Precise fluid replacement was administrated consistent with the standard administration guidelines during anaesthesia.
* Patients were ventilated using Datex-Ohmeda Aestiva/5 (Madison, WI) anaesthesia machine, (volume controlled mode) with lung protective strategy using a tidal volume of 6- 8 ml/kg ideal body weight, (5-10 cm H20) PEEP and 50 % O2 in air adjusted to reach Spo2 ≥ 95 %. The respiratory rate was adjusted to keep end - tidal Co2 level between (35 -45 mmHg), and inspiratory to expiratory times at a ratio 1:2.
* Measurements

  1. Hemodynamic parameters: HR and MAP.
  2. Respiratory mechanics: Peak airway pressure (Paw-peak) and Plateau pressure (Paw-plat).
  3. Oxygenation parameters: Partial arterial tension of oxygen (PaO2), PaO2/FiO2 ratio and oxygen saturation (SpO2).

     All the previous measurements were recorded at the following time points: T0 (baseline value on room air), T5 (5 minutes after pneumoperitoneum), T30 (30 minutes after first RM), T6o (60 minutes after first RM), T90 (90 minutes after first RM), TE (20 minutes after the end of surgery on nasal cannula 3 L /min). Additional arterial blood gases analysis was performed in the PACU after 30 mins and 1 hr postoperatively.
  4. Serum interleukins (IL)-6 and (IL)-8, using enzyme-linked immunosorbent assay (ELISA) (Biosource, Biosite, Germany) in (pg/ml) were measured as baseline preoperative value and after 24 hr postoperatively. Validation of methods and degrees of concentrations was done following to the accompanied instructions.
  5. Postoperative pulmonary and non-pulmonary complication - (if any) - were assessed and reported in the PACU.
  6. Other variables like: duration of anaesthesia, duration of surgery, pneumoperitoneum time, number of patients needed vasopressors, length of ICU stay and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

- American Society of Anaesthesiologists physical Status classification scores of 1-2, scheduled for laparoscopic bariatric procedures

Exclusion Criteria:

* patients refusal,
* history of significant pulmonary disease (obstructive or restrictive),
* previous pneumothorax,
* significant cardiac dysfunction (arrhythmias ± unstable haemodynamics
* left ventricular ejection fraction < 40%)
* difficult intubation
* significant hepatic or renal impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-05 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Partial arterial tension of oxygen (PaO2), | 20 minutes postoperatively
Serum interleukins (IL)-6 | after 24 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University Faculty of Medicin, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No